CLINICAL TRIAL: NCT04688957
Title: Osseodensification by Densah Burs Versus Osteotome for Transcrestal Maxillary Sinus Lifting With Simultaneous Implant Placement (Randomized Clinical Trial)
Brief Title: Osseodensification by Densah Burs Versus Osteotome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: osseodensifcation
Record Dates: First submitted 2020-12-18; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Maxillary Sinus Lift

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- osteotome sinus lifting (Active Comparator)
  Interventions: Procedure: osteotome sinus lifting
- oseodensification sinus lifting (Experimental)
  Interventions: Procedure: oseodensification sinus lifting

INTERVENTIONS:
Procedure: oseodensification sinus lifting — application of first densah bur with densifying mood (reverse) counterclockwise, 1200 revolution per minute until the sinus is reached then use a wider densah bur with the same mode and bouncing motion to elevate the sinus floor up to 3 mm in 1mm increments.
  Arms: oseodensification sinus lifting
Procedure: osteotome sinus lifting — drilling implant site with consecutive drills short of the sinus floor by 1-2mm , using osteotome in appropriate size and application of one tap until sinus floor is elevated, using the final drill for the desired implant diameter
  Arms: osteotome sinus lifting

SUMMARY:
implant placement in the posterior maxilla is problematic, not only due to inferior properties of bone but also due to loss of vertical bone height which happens after extraction of posterior teeth. when the required additional height is few millimeters, indirect transcresta sinus lifting procedures are recommended.

This study compares sinus lifting using the conventional osteotome versus the osseodensification with densah burs.

DETAILED DESCRIPTION:
a total of 12 patients with missing maxillary premolars or molars and with limited vertical bone height below the maxillary sinus floor will receive implants either with osteotome or with Densah burs transcrestal sinus lifting to compare clinically and radiographically transcrestal sinus lifting with Densah burs and osteotome with simultaneous implant placement

ELIGIBILITY:
Inclusion Criteria:

* Patient with missing maxillary premolas and molars
* Vertical bone height of 5-8 mm
* Non smokers
* Good oral hygiene

Exclusion Criteria:

* Bad oral hygiene
* maxillary sinusitis
* Presence of infection or periapical lesions in adjacent teeth
* Bruxism or clenching
* Alcoholism
* Medically compromised patients with a condition that affect the procedure
* Multiple sinus septa

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
implant stability | at 6 months
  Using the Osstell, The result is presented as an ISQ value of 1-100. The higher the ISQ, the more stable the implant
change in bone height | at baseline and 6 months
  using CBCT
change in bone density | at baseline and 6 months
  using CBCT

SECONDARY OUTCOMES:
Pain scores | at 2 weeks
  10-point Visual Analogue Scale (VAS). (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
edema scores | at 2 weeks
  The pitting is graded on a scale of +1 to +4 as follows:
  * +1 (trace) slight indentation rapid return to normal.
  * +2 (mild) the indentation returns to normal in a few seconds.
  * +3 (moderate) 6 mm indentation rebounds in 10-20 seconds.
  * +4 (severe) 8 mm indentation rebounds in more than 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Elghobashy MTM, Shaaban AM, Melek LNF. Radiographic comparison between Densah burs and osteotome for graftless internal sinus lifting with simultaneous implant placement: a randomized clinical trial. Int J Oral Maxillofac Surg. 2023 Mar;52(3):388-395. doi: 10.1016/j.ijom.2022.06.020. Epub 2022 Jul 13. PMID 35840446